CLINICAL TRIAL: NCT00005131
Title: Atherosclerosis Risk in Communities (ARIC)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1001
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Atherosclerosis; Coronary Disease; Coronary Heart Disease Risk Reduction; Diabetes Mellitus; Cardiovascular Diseases; Heart Diseases; Heart Failure, Congestive; Heart Failure
MeSH Terms: conditions — Atherosclerosis; Coronary Disease; Diabetes Mellitus; Cardiovascular Diseases; Heart Diseases; Heart Failure

SUMMARY:
To measure associations of established and suspected coronary heart disease risk factors with both atherosclerosis and new coronary heart disease events in representative cohorts from four diverse United States communities. To compare the communities with respect to risk factors, medical care, atherosclerosis, and coronary heart disease incidence. ARIC has two components in each community: study of representative cohorts of adult men and women, and community surveillance of morbidity and mortality.

DETAILED DESCRIPTION:
BACKGROUND:

Although it is now firmly established that coronary heart disease mortality rates in the United States have fallen by about 50 percent since the mid 1960's, there has been no systematic program to study in parallel coronary heart disease morbidity and the prevalence of atherosclerosis. Such information is essential for an understanding of the factors influencing the time trends, for quantifying the effects of prevention versus treatment, and for guiding future policy in research and services. It remains a possibility that the mortality decline in past years was not accompanied by a reduction in incidence, or a diminution in the extent of the underlying arterial diseases. A trend confined to mortality would require different explanations and call for different strategies of prevention than a decline encompassing the whole spectrum of clinical manifestations, which would favor a risk factor explanation. ARIC surveillance provides cardiovascular incidence rates, and its cohorts provide information on atherosclerosis, cardiovascular symptoms, new and established risk factors and medical care utilization on representative residents of each community. New predictors of both atherosclerosis and cardiovascular diseases are investigated using data obtained at four examination centers, the ultrasound center and five central laboratories.

The 1978 Conference on the Decline in Coronary Heart Disease Mortality and the 1979 Working Group on Heart Disease Epidemiology both recommended a community surveillance program. As a result, in 1980 the Clinical Applications and Prevention Advisory Committee and the National Heart, Lung, and Blood Advisory Council approved Phase I of the surveillance pilot study. Phase II of the pilot study and the full-scale study was approved by the Clinical Applications and Prevention Advisory Committee in May 1982. The Requests for Proposals for ARIC were released in September 1984 and awards made in 1985.

DESIGN NARRATIVE:

ARIC is a large-scale, long-term program that measures associations of established and suspected CHD risk factors with both atherosclerosis and new CHD events in men and women from four diverse communities. The project has two components: community surveillance of morbidity and mortality, and repeated examinations of a representative cohort of men and women in each community. The representative cohorts include 4,000 persons from each community. Three of these reflect the ethnic composition of the communities in which they live; one cohort is black. The community surveillance involves abstracting hospital records and death certificates and investigating out-of-hospital deaths for hospitalized myocardial infarction and CHD death in 800,000 men and women in these four communities.

All cohort participants were examined four times (1987-90, and 1990-93, 1993-96, and 1996-99), and were contacted annually to update their medical histories. Atherosclerosis was measured by carotid ultrasonography. Arteriosclerosis was measured using retinal photography. Cerebrovascular disease was assessed using MRI in a sample of black and white participants. Risk factors studied include: blood lipids, lipoprotein cholesterols, and apolipoproteins; plasma hemostatic factors; blood chemistries and hematology and indicators of infectious and inflammatory disease; DNA markers of these risk factors, sitting, supine and standing blood pressures; anthropometry; fasting blood glucose and insulin levels; ECG findings; heart rate variability; cigarette and alcohol use; physical activity levels; dietary aspects; and family history. Novel factors are tested using nested case-control studies on stored blood.

The fourth and final examination, which included a complete periodontal examination with measures of inflammatory markers was completed in 1999, with a return rate of 86%. Community surveillance currently provides complete age, race, and sex-specific rates of hospitalization for myocardial infarction and coronary heart disease death in the communities for 1987-1997.

The study has been extended through January, 2007 to continue to follow the cohort through annual telephone calls and hospital surveillance to identify incident cardiovascular events through 19 years. Community surveillance continues to identify trends in cardiovascular disease incidence, case-fatality, and mortality in 35-74 year olds over a 19 year period.

The diverse communities can be compared with respect to CHD incidence and medical care and, through the cohort component, with respect to risk factors and peripheral atherosclerosis. The results will provide a measure of the variation in the distribution and determinants of CHD in the U.S. and, within the limits of ecologic analysis, suggest possible reasons for observed differences.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christie Ballantyne — Baylor College of Medicine; Lloyd Chambless — University of North Carolina; Josef Coresh — Johns Hopkins University; Matthew Davis — University of Wisconsin, Madison; Aaron Folsom — University of Minnesota; Gerardo Heiss — University of North Carolina; Daniel Jones — University of Mississippi Medical Center; Kenneth Wu — Texas Health Science Center

REFERENCES:
- [Background] Please refer to the ARIC website for the complete bibliography: http://www.bios.unc.edu/cscc/ARIC/
- [Derived] Tong Y, Jia Y, Gong A, Li F, Zeng R. Systemic inflammation in midlife is associated with late-life functional limitations. Sci Rep. 2024 Jul 29;14(1):17434. doi: 10.1038/s41598-024-68724-w. PMID 39075139
- [Derived] Li Y, Jia Y, Jiang W, Li D, Yu J, Liu Y, Liao X, Zhao Z. Association between cognitive impairment and risk of atrial fibrillation: The Atherosclerosis Risk in Communities study. Cardiol J. 2024;31(4):553-563. doi: 10.5603/cj.93107. Epub 2023 Oct 19. PMID 37853826
- [Derived] Jia Y, Li D, Yu J, Liu Y, Li F, Li W, Zhang Q, Gao Y, Zhang W, Zeng Z, Zeng R, Liao X, Zhao Q, Wan Z. Subclinical cardiovascular disease and frailty risk: the atherosclerosis risk in communities study. BMC Geriatr. 2022 Apr 12;22(1):321. doi: 10.1186/s12877-022-02974-z. PMID 35413794
- [Derived] Zhuang XD, Tian T, Liao LZ, Dong YH, Zhou HJ, Zhang SZ, Chen WY, Du ZM, Wang XQ, Liao XX. Deep Phenotyping and Prediction of Long-term Cardiovascular Disease: Optimized by Machine Learning. Can J Cardiol. 2022 Jun;38(6):774-782. doi: 10.1016/j.cjca.2022.02.008. Epub 2022 Feb 11. PMID 35157988
- [Derived] Arora S, Brown ZD, Sivaraj K, Hendrickson MJ, Mazzella AJ, Chang PP, Vaduganathan M, Qamar A, Gehi AK, Pandey A, Vavalle JP. The Relationship Between Atrial Fibrillation, Mitral Regurgitation, and Heart Failure Subtype: The ARIC Study. J Card Fail. 2022 Jun;28(6):883-892. doi: 10.1016/j.cardfail.2021.10.015. Epub 2021 Dec 23. PMID 34955335
- [Derived] Li D, Jia Y, Yu J, Liu Y, Li F, Liu Y, Wu Q, Liao X, Zeng Z, Zeng R, Wan Z. Adherence to Healthy Lifestyle and the Risk of Function Limitations in Late Life: The Atherosclerosis Risk in Communities Study. Front Aging Neurosci. 2021 Aug 3;13:698699. doi: 10.3389/fnagi.2021.698699. eCollection 2021. PMID 34413768
- [Derived] Li D, Jia Y, Yu J, Liu Y, Li F, Liu Y, Wu Q, Liao X, Zeng Z, Wan Z, Zeng R. Adherence to a Healthy Lifestyle and the Risk of All-Cause Mortality and Cardiovascular Events in Individuals With Diabetes: The ARIC Study. Front Nutr. 2021 Jul 5;8:698608. doi: 10.3389/fnut.2021.698608. eCollection 2021. PMID 34291073
- [Derived] Li F, Li D, Yu J, Jia Y, Liu Y, Liu Y, Wu Q, Liao X, Zeng Z, Wan Z, Zeng R. Silent Myocardial Infarction and Long-Term Risk of Frailty: The Atherosclerosis Risk in Communities Study. Clin Interv Aging. 2021 Jun 18;16:1139-1149. doi: 10.2147/CIA.S315837. eCollection 2021. PMID 34168437
- [Derived] Gao JW, Hao QY, Gao M, Zhang K, Li XZ, Wang JF, Vuitton DA, Zhang SL, Liu PM. Triglyceride-glucose index in the development of peripheral artery disease: findings from the Atherosclerosis Risk in Communities (ARIC) Study. Cardiovasc Diabetol. 2021 Jun 24;20(1):126. doi: 10.1186/s12933-021-01319-1. PMID 34167539
- [Derived] Sun XT, Zeng C, Zhang SZ, Zhou HM, Zhong XB, Xiong ZY, Yang DY, Guo Y, Zhuang XD, Liao XX. Long-term tracking of fasting blood glucose variability and peripheral artery disease in people without diabetes. BMJ Open Diabetes Res Care. 2020 Sep;8(1):e000896. doi: 10.1136/bmjdrc-2019-000896. PMID 32994225
- [Derived] DeBarmore B, Longchamps RJ, Zhang Y, Kalyani RR, Guallar E, Arking DE, Selvin E, Young JH. Mitochondrial DNA copy number and diabetes: the Atherosclerosis Risk in Communities (ARIC) study. BMJ Open Diabetes Res Care. 2020 Aug;8(1):e001204. doi: 10.1136/bmjdrc-2020-001204. PMID 32801120
- [Derived] Fashanu OE, Zhao D, Schneider ALC, Rawlings AM, Sharrett AR, Lutsey PL, Gottesman RF, Gross AL, Guallar E, Alonso A, Mosley TH, Michos ED. Mid-life serum Vitamin D concentrations were associated with incident dementia but not late-life neuropsychological performance in the Atherosclerosis Risk in Communities (ARIC) Study. BMC Neurol. 2019 Oct 22;19(1):244. doi: 10.1186/s12883-019-1483-3. PMID 31640594
- [Derived] Thorvaldsen T, Claggett BL, Shah A, Cheng S, Agarwal SK, Wruck LM, Chang PP, Rosamond WD, Lewis EF, Desai AS, Lund LH, Solomon SD. Predicting Risk in Patients Hospitalized for Acute Decompensated Heart Failure and Preserved Ejection Fraction: The Atherosclerosis Risk in Communities Study Heart Failure Community Surveillance. Circ Heart Fail. 2017 Dec;10(12):e003992. doi: 10.1161/CIRCHEARTFAILURE.117.003992. PMID 29242352
- [Derived] McKeown NM, Dashti HS, Ma J, Haslam DE, Kiefte-de Jong JC, Smith CE, Tanaka T, Graff M, Lemaitre RN, Rybin D, Sonestedt E, Frazier-Wood AC, Mook-Kanamori DO, Li Y, Wang CA, Leermakers ETM, Mikkila V, Young KL, Mukamal KJ, Cupples LA, Schulz CA, Chen TA, Li-Gao R, Huang T, Oddy WH, Raitakari O, Rice K, Meigs JB, Ericson U, Steffen LM, Rosendaal FR, Hofman A, Kahonen M, Psaty BM, Brunkwall L, Uitterlinden AG, Viikari J, Siscovick DS, Seppala I, North KE, Mozaffarian D, Dupuis J, Orho-Melander M, Rich SS, de Mutsert R, Qi L, Pennell CE, Franco OH, Lehtimaki T, Herman MA. Sugar-sweetened beverage intake associations with fasting glucose and insulin concentrations are not modified by selected genetic variants in a ChREBP-FGF21 pathway: a meta-analysis. Diabetologia. 2018 Feb;61(2):317-330. doi: 10.1007/s00125-017-4475-0. Epub 2017 Nov 2. PMID 29098321
- [Derived] Ogilvie RP, Lutsey PL, Heiss G, Folsom AR, Steffen LM. Dietary intake and peripheral arterial disease incidence in middle-aged adults: the Atherosclerosis Risk in Communities (ARIC) Study. Am J Clin Nutr. 2017 Mar;105(3):651-659. doi: 10.3945/ajcn.116.137497. Epub 2017 Jan 11. PMID 28077376
- [Derived] Pokharel Y, Sun W, Virani SS, Nambi V, Hoogeveen RC, Chang PP, Ndumele CE, Solomon SD, Bozkurt B, Selvin E, Ballantyne CM, Deswal A. Myocardial Injury, Obesity, and the Obesity Paradox: The ARIC Study. JACC Heart Fail. 2017 Jan;5(1):56-63. doi: 10.1016/j.jchf.2016.10.010. Epub 2016 Dec 21. PMID 28017350
- [Derived] Tanaka T, Ngwa JS, van Rooij FJ, Zillikens MC, Wojczynski MK, Frazier-Wood AC, Houston DK, Kanoni S, Lemaitre RN, Luan J, Mikkila V, Renstrom F, Sonestedt E, Zhao JH, Chu AY, Qi L, Chasman DI, de Oliveira Otto MC, Dhurandhar EJ, Feitosa MF, Johansson I, Khaw KT, Lohman KK, Manichaikul A, McKeown NM, Mozaffarian D, Singleton A, Stirrups K, Viikari J, Ye Z, Bandinelli S, Barroso I, Deloukas P, Forouhi NG, Hofman A, Liu Y, Lyytikainen LP, North KE, Dimitriou M, Hallmans G, Kahonen M, Langenberg C, Ordovas JM, Uitterlinden AG, Hu FB, Kalafati IP, Raitakari O, Franco OH, Johnson A, Emilsson V, Schrack JA, Semba RD, Siscovick DS, Arnett DK, Borecki IB, Franks PW, Kritchevsky SB, Lehtimaki T, Loos RJ, Orho-Melander M, Rotter JI, Wareham NJ, Witteman JC, Ferrucci L, Dedoussis G, Cupples LA, Nettleton JA. Genome-wide meta-analysis of observational studies shows common genetic variants associated with macronutrient intake. Am J Clin Nutr. 2013 Jun;97(6):1395-402. doi: 10.3945/ajcn.112.052183. Epub 2013 May 1. PMID 23636237
- [Derived] Yang EY, Chambless L, Sharrett AR, Virani SS, Liu X, Tang Z, Boerwinkle E, Ballantyne CM, Nambi V. Carotid arterial wall characteristics are associated with incident ischemic stroke but not coronary heart disease in the Atherosclerosis Risk in Communities (ARIC) study. Stroke. 2012 Jan;43(1):103-8. doi: 10.1161/STROKEAHA.111.626200. Epub 2011 Oct 27. PMID 22033999
- [Derived] Chatterjee R, Yeh HC, Shafi T, Anderson C, Pankow JS, Miller ER, Levine D, Selvin E, Brancati FL. Serum potassium and the racial disparity in diabetes risk: the Atherosclerosis Risk in Communities (ARIC) Study. Am J Clin Nutr. 2011 May;93(5):1087-91. doi: 10.3945/ajcn.110.007286. Epub 2011 Mar 2. PMID 21367942
- [Derived] Yang EY, Nambi V, Tang Z, Virani SS, Boerwinkle E, Hoogeveen RC, Astor BC, Mosley TH, Coresh J, Chambless L, Ballantyne CM. Clinical implications of JUPITER (Justification for the Use of statins in Prevention: an Intervention Trial Evaluating Rosuvastatin) in a U.S. population insights from the ARIC (Atherosclerosis Risk in Communities) study. J Am Coll Cardiol. 2009 Dec 15;54(25):2388-95. doi: 10.1016/j.jacc.2009.10.006. PMID 20082929
- [Derived] Myerson M, Coady S, Taylor H, Rosamond WD, Goff DC Jr; ARIC Investigators. Declining severity of myocardial infarction from 1987 to 2002: the Atherosclerosis Risk in Communities (ARIC) Study. Circulation. 2009 Feb 3;119(4):503-14. doi: 10.1161/CIRCULATIONAHA.107.693879. Epub 2009 Jan 19. PMID 19153274
- See also: Related Info — http://www.cscc.unc.edu/aric/
- Available data/document: Individual Participant Data Set: ARIC — http://biolincc.nhlbi.nih.gov/studies/aric/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Forms — http://www2.cscc.unc.edu/aric/cohort-forms
- Available data/document: Study Manuals — http://www2.cscc.unc.edu/aric/cohort-forms